CLINICAL TRIAL: NCT00158119
Title: Ameliorating Disability Through Power Training
Brief Title: A Comparison of Weighted Vest Exercise and Strength Training
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Spaulding Rehabilitation Hospital PM&R (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0037; K23AG019663-01 (NIH)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Mobility Limitations; Aging
Keywords: strength training; power training; exercise training; functional performance tasks
MeSH Terms: conditions — Mobility Limitation

INTERVENTIONS:
Behavioral: InVEST (Increased Velocity Exercise Specific to Task)

SUMMARY:
The purpose of this study is to evaluate two types of exercise therapy designed to improve muscle power and mobility: weighted vest exercise vs. progressive resistance training.

DETAILED DESCRIPTION:
Muscle power, a separate physical attribute from strength, is an important determinate of physical functioning in the elderly, for example in avoiding impending falls, rising from a chair, and climbing stairs. Muscle power, which declines with aging at a different rate than strength, has been shown in previous studies to improve through power training utilizing specially designed exercise equipment. However, weighted vest exercise could provide an acceptable, low cost, readily accessible alternative.

The hypotheses being tested in this study are: 1) weighted vest exercise will improve lower extremity power when compared to age matched controls in a standardized progressive resistance training program; 2) improvements in lower extremity power enhance functional performance as shown by improved gait velocity, stair climbing, and chair rise time; and 3) weighted vest exercise in impaired older adults will improve self-reported function and disability.

One hundred sixty-four men and women ages 65 and older, with some physical limitation but able to climb stairs independently, will be randomized to one of two 16-week exercise programs. The intervention group will participate in a weighted vest exercise protocol, consisting of chair-based and stair-climbing exercise, while the control group will participate in a standardized progressive resistance training program. Participants in both programs will meet three times per week for 30-60 minutes per session, for a total of 16 weeks, at a research exercise gym, and will be under the direct supervision of research staff.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling men and women aged 65 or older
* Ability to provide informed consent
* Impairment in physical performance, based on a score between 4 and 10 inclusive on the SPPB (Short Physical Performance Battery), which evaluates standing balance, walking speed, and chair-rise time
* Score of 24 or greater on the Folstein mini-mental status exam
* Exhibit independent stair-climbing ability

Exclusion Criteria:

* Unstable acute or chronic disease
* Neuromusculoskeletal impairment interfering with independent stair climbing
* Abdominal aortic aneurysm
* Exertional angina
* History of ventricular arrhythmia
* Inguinal or abdominal hernia
* Symptomatic valvular heart disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160
Dates: Start 2001-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Leg power
leg strength
mobility
endurance
balance measured at baseline, 8 weeks, and 16 weeks

SECONDARY OUTCOMES:
Disability

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan F. Bean, MD, MS, Principal Investigator — Spaulding Cambridge Outpatient Center
Locations (1):
- Spaulding Cambridge Outpatient Center, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Bean JF, Kiely DK, Herman S, Leveille SG, Mizer K, Frontera WR, Fielding RA. The relationship between leg power and physical performance in mobility-limited older people. J Am Geriatr Soc. 2002 Mar;50(3):461-7. doi: 10.1046/j.1532-5415.2002.50111.x. PMID 11943041
- [Background] Bean J, Herman S, Kiely DK, Callahan D, Mizer K, Frontera WR, Fielding RA. Weighted stair climbing in mobility-limited older people: a pilot study. J Am Geriatr Soc. 2002 Apr;50(4):663-70. doi: 10.1046/j.1532-5415.2002.50160.x. PMID 11982666
- [Background] Fielding RA, LeBrasseur NK, Cuoco A, Bean J, Mizer K, Fiatarone Singh MA. High-velocity resistance training increases skeletal muscle peak power in older women. J Am Geriatr Soc. 2002 Apr;50(4):655-62. doi: 10.1046/j.1532-5415.2002.50159.x. PMID 11982665
- [Background] Bean JF, Herman S, Kiely DK, Frey IC, Leveille SG, Fielding RA, Frontera WR. Increased Velocity Exercise Specific to Task (InVEST) training: a pilot study exploring effects on leg power, balance, and mobility in community-dwelling older women. J Am Geriatr Soc. 2004 May;52(5):799-804. doi: 10.1111/j.1532-5415.2004.52222.x. PMID 15086665
- [Background] Bean JF, Vora A, Frontera WR. Benefits of exercise for community-dwelling older adults. Arch Phys Med Rehabil. 2004 Jul;85(7 Suppl 3):S31-42; quiz S43-4. doi: 10.1016/j.apmr.2004.03.010. PMID 15221722
- [Derived] Li X, Forman DE, Kiely DK, LaRose S, Hirschberg R, Frontera WR, Bean JF. Validity of an exercise test based on habitual gait speed in mobility-limited older adults. Arch Phys Med Rehabil. 2012 Feb;93(2):344-50. doi: 10.1016/j.apmr.2011.08.032. PMID 22289248
- [Derived] Suri P, Kiely DK, Leveille SG, Frontera WR, Bean JF. Increased trunk extension endurance is associated with meaningful improvement in balance among older adults with mobility problems. Arch Phys Med Rehabil. 2011 Jul;92(7):1038-43. doi: 10.1016/j.apmr.2010.12.044. Epub 2011 Jun 2. PMID 21636073
- [Derived] Bean JF, Kiely DK, LaRose S, Goldstein R, Frontera WR, Leveille SG. Are changes in leg power responsible for clinically meaningful improvements in mobility in older adults? J Am Geriatr Soc. 2010 Dec;58(12):2363-8. doi: 10.1111/j.1532-5415.2010.03155.x. PMID 21143443
- [Derived] Suri P, Kiely DK, Leveille SG, Frontera WR, Bean JF. Trunk muscle attributes are associated with balance and mobility in older adults: a pilot study. PM R. 2009 Oct;1(10):916-24. doi: 10.1016/j.pmrj.2009.09.009. PMID 19854420
- [Derived] Bean JF, Kiely DK, LaRose S, O'Neill E, Goldstein R, Frontera WR. Increased velocity exercise specific to task training versus the National Institute on Aging's strength training program: changes in limb power and mobility. J Gerontol A Biol Sci Med Sci. 2009 Sep;64(9):983-91. doi: 10.1093/gerona/glp056. Epub 2009 May 4. PMID 19414509